CLINICAL TRIAL: NCT01357811
Title: A Single-site, Open-label, Fixed-sequence Phase 1 Study Evaluating the Effect of Eliglustat (Genz-112638) on the Pharmacokinetics and Safety and Tolerability of Digoxin in Healthy Adult Subjects
Brief Title: A Phase 1 Study Evaluating Eliglustat's Effects on Pharmacokinetics, Safety & Tolerability of Digoxin in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: GZGD03610
Record Dates: First submitted 2011-05-19; First posted 2011-05-23 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Healthy Volunteer
Keywords: Genz-112638; digoxin
MeSH Terms: interventions — eliglustat; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- digoxin (Active Comparator)
  Interventions: Drug: digoxin
- eliglustat with digoxin (Experimental)
  Interventions: Drug: eliglustat; digoxin

INTERVENTIONS:
Drug: eliglustat; digoxin — repeat oral doses of 150 mg BID (or 100 mg BID if a CYP2D6 poor metabolizer) eliglustat (Day 11 to Day 17) plus singe dose of digoxin 0.25mg on Day 15
  Other Names: Genz-112638
  Arms: eliglustat with digoxin
Drug: digoxin — oral 0.25mg dose of digoxin (single dose) on Day 1
  Arms: digoxin

SUMMARY:
The primary objective of this study is to determine the effect of repeat oral doses of eliglustat 150 mg twice daily (BID) (or 100 mg BID for CYP2D6 poor metabolizers) on the pharmacokinetics (PK) of orally administered digoxin 0.25 mg in healthy adult subjects. This will be a single-site, open-label study in 2 staggered cohorts of healthy adult subjects. The study will comprise a screening period (between Day -45 and Day -2), treatment period 1 (Day -1 to Day 4), treatment period 2 (Day 11 to Day 18), and a safety follow-up visit (Day 24 ± 1). There will be a 10-day washout between dosing of study drug in Period 1 and Period 2. The duration of each subject's participation in the study, inclusive of the screening and follow-up visits, will be approximately 10 weeks.

DETAILED DESCRIPTION:
Cohort 1 will comprise 10 subjects and Cohort 2 will comprise 18 subjects. Initiation of treatment in Cohort 1 will occur at least 6 days prior to the start of treatment for Cohort 2. In each cohort, eligible subjects will be admitted to the clinical facility on Day -1, the day prior to the start of dosing in Period 1, and will remain in the clinic until completion of study procedures on Day 18, the last day of Period 2 (an approximately 18-night inpatient stay). In Period 1, all subjects will receive a single oral dose of digoxin 0.25 mg on Day 1. In Period 2, subjects will receive repeat oral doses of eliglustat 150 mg BID (or 100 mg BID if a CYP2D6 poor metabolizer) from Day 11 to Day 17 and a single oral dose of digoxin 0AA mg on Day 15. For Cohort 2, co-administration of digoxin and eliglustat on Day 15 will occur only after review of safety data (including telemetry data) through at least Day 16 for all subjects in Cohort 1. The decision to proceed with concomitant dosing of subjects in Cohort 2 will be at the discretion of the Investigator, with consultation of the Sponsor, as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* The male or female subject is in good general health
* The subject has a body weight of 50 to 100 kg (110 to 220 lb) with a body mass index (BMI) ≤32 kg/m2 at screening.
* The subject's physical examination, laboratory, vital sign, and electrocardiogram (ECG) test results are within normal limits at screening and Day -1 or, if abnormal, are not considered clinically significant in the opinion of the Investigator.
* The subject has been a non-smoker for at least 6 months prior to the time of providing informed consent, and is willing and able to abstain from smoking (and use of other forms of nicotine) until completion of the safety follow-up visit.
* The subject has not used drugs of abuse for at least 6 months prior to Day -1 and is willing and able to abstain from using drugs of abuse until completion of the safety follow-up visit.
* The subject is willing and able to abstain from alcohol for 48 hours prior to the first dose of study drug until completion of the safety follow-up visit.
* The subject is willing and able to abstain from grapefruit and grapefruit juice for 72 hours prior to the first dose of study drug until completion of the safety follow-up visit.
* The subject is willing and able to maintain a normal-fiber diet (i.e., to abstain from excess fiber-rich foods) for 72 hours prior to the first dose of study drug until completion of the safety follow-up visit.
* Female subjects of childbearing potential must have a documented negative pregnancy test at screening and Day 1, and be willing to use a medically accepted form of contraception (as defined in the protocol) from screening until 30 days after the last dose of study drug. A woman of childbearing potential is defined as any female who has not been amenorrheic for at least 2 years or has not undergone a hysterectomy or surgical sterilization.

Exclusion Criteria:

* The subject has any of the following: Clinically significant coronary artery disease including history of myocardial infarction or ongoing signs or symptoms consistent with cardiac ischemia or heart failure; clinically significant arrhythmias or conduction defect such as 2nd or 3rd degree atrioventricular (AV) block, a PR interval ≥210 msec, complete bundle branch block, prolonged QTc interval (e.g., repeated demonstration of a QTc interval ≥450 msec), or sustained ventricular tachycardia.
* The subject has received antibiotics for any reason within 30 days prior to the first dose of study drug.
* The subject has received any other prescription or non-prescription medication (with the exception of nonprescription-strength ibuprofen and acetaminophen) or dietary or herbal or fiber supplement within 30 days or 5 half-lives (whichever is longer) prior to the first dose of study drug without the approval of the Investigator and Genzyme.
* The subject receives an immunization within 30 days of providing informed consent.
* The subject has a history of hypersensitivity to digoxin or other digitalis glycosides, or has other drug allergies that are clinically significant in the opinion of the Investigator (e.g., significant rash or hives).
* The subject has a clinically significant organic disease, including cardiovascular, renal, hepatic, gastrointestinal, pulmonary, neurologic, endocrine, metabolic, or psychiatric disease, or other medical condition such as electrolyte disorders, serious intercurrent illness, or extenuating circumstance that, in the opinion of the Investigator, precludes participation in the trial.
* The subject has digestive disorders, including malabsorption, gastroenteritis, pancreatitis, constipation, gastroesophageal reflux disease, diverticulitis, irritable bowel syndrome, or inflammatory bowel disease (including Crohn's disease).
* The subject has had a cholecystectomy.
* The subject has a screening laboratory test result >2x the upper limit of normal (ULN) for any of the following liver function tests: aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma glutamyltransferase (GGT), and total bilirubin.
* The subject tests positive for human immunodeficiency virus (HIV) antibody, hepatitis C antibody, or hepatitis B surface antigen at screening.
* The subject tests positive for urine drugs of abuse, urine alcohol, or urine cotinine at screening.
* The subject received an investigational product within 30 days prior to providing informed consent or plans to receive any other investigational product at any time during the course of this study.
* The subject donated blood or blood products within 30 days prior to providing informed consent.
* The subject's schedule or travel plans prevent the completion of all required visits.
* The subject is scheduled for inpatient hospitalization, including elective surgery (inpatient or outpatient), during the study.
* The subject has a history of cancer, with the exception of basal cell carcinoma.
* The female subject of childbearing potential is pregnant or lactating.
* The subject, in the opinion of the Investigator, is unable to adhere to the requirements of the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2011-08; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics as measured by area under the serum concentration time curve (AUC) of digoxin alone and in combination with eliglustat | 18 days
Pharmacokinetics as measured by maximum serum concentration (Cmax) following administration of digoxin alone and in combination with eliglustat | 18 days

SECONDARY OUTCOMES:
Pharmacokinetics for digoxin as measured by the time to maximum serum concentration (Tmax) following administration of digoxin alone and in combination with eliglustat | 18 days
Pharmacokinetics for digoxin as measured by terminal elimination half-life (T1/2) following administration of digoxin alone and in combination with eliglustat | 18 days
Pharmacokinetics for digoxin as measured by apparent serum clearance (CL) following administration of digoxin alone and in combination with eliglustat | 18 days
Pharmacokinetics for digoxin as measured by renal clearance (CLr) following administration of digoxin alone and in combination with eliglustat | 18 days
Pharmacokinetics as measured by amount of digoxin excreted in the urine over 72 hours (Ae) following administration of digoxin alone and in combination with eliglustat. | 18 days
Pharmacokinetics as measured by eliglustat trough concentrations following administration of digoxin in combination with eliglustat | 18 days
Safety as measured by the incidence, seriousness and severity of adverse events (AEs). | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (1):
- PPD Phase I Clinic, Austin, Texas, United States